CLINICAL TRIAL: NCT03799120
Title: The Effect of Daily Versus Twice Per Day Tamsulosin on Ureteral Stent Symptoms Following Ureteroscopy for Nephrolithiasis
Brief Title: Daily Versus Twice Per Day Tamsulosin for Ureteral Stent Symptoms
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Gundersen Lutheran Medical Foundation (Other)
Responsible Party: Principal Investigator, Kara Kallies, Academic Researcher / study coordinator, Gundersen Lutheran Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2-18-11-001
Record Dates: First submitted 2019-01-04; First posted 2019-01-10 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Ureteral Diseases
MeSH Terms: conditions — Ureteral Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- tamsulosin QD + Placebo (Placebo Comparator): 0.4 mg tamsulosin QD + Placebo QD
  Interventions: Drug: Tamsulosin BID; Other: Placebo
- tamsulosin BID (Experimental): 0.4 mg tamsulosin BID
  Interventions: Drug: Tamsulosin BID

INTERVENTIONS:
Drug: Tamsulosin BID — comparison of once daily versus twice daily tamsulosin
Other: Placebo — Placebo
  Arms: tamsulosin QD + Placebo

SUMMARY:
A single-center prospective, randomized study to assess two different dosing regimens (0.4 mg QD vs. 0.4 mg BID) of tamsulosin for ureteral stent-related discomfort will be completed.

DETAILED DESCRIPTION:
Ureteral stents are commonly used to maintain patency of the ureter and are placed for several common reasons including ureteral obstruction due to nephrolithiasis, cancer, or fibrosis as well as after surgical interventions involving ureteroscopy, ureteral anastomoses or prophylactically prior to extracorporeal shock wave lithotripsy. Ureteral stents have been associated with significant discomfort and dissatisfaction among patients.5 Bosio and colleagues noted that among patients with indwelling stents, 59.1% reported daily urinary frequency ≥ 1 per hour, 90.1% reported ≥ 1 nocturnal micturition episodes, 86.6% reported urinary urgency, and 82.3% reported dysuria. Further, 83.2% complained of pain, mostly in the kidney (67.9%) or in the bladder area (31.3%), particularly during physical activity. Over 90% of patients reported that this pain interfered with their everyday life.

The Ureteric Stent Symptom Questionnaire (USSQ) was developed in 2003 by Joshi and colleagues to quantify patients' discomfort relating specifically to ureteral stents. The USSQ measures several domains relating to stent pain including general health, urinary issues, pain, work performance, sexual matters, and quality of life with stent in situ. The USSQ has been validated and translated and is currently a widely used measure.

While commonly used for treatment of benign prostatic hyperplasia, several studies have evaluated the efficacy of α-blockers for stent pain and have demonstrated a significant improvement in USSQ scores using α-blockers (mean reduction of 8.4 in urinary symptom scores and 7.2 in body pain scores). To date, randomized controlled trials have used one of two types of α-blockers: tamsulosin (0.4mg) vs. alfuzosin (10 mg). In treating benign prostatic hyperplasia, a total maximum dose of 0.8mg tamsulosin is used (either 0.4mg BID or 0.8mg daily), which has shown increased efficacy compared to the 0.4mg QD dose without an increase in adverse effects. Currently, tamsulosin 0.4mg daily is the off-label dosage indicated for lower urinary tract symptoms for patients with an indwelling stent. No study to date, however, has evaluated the clinical impact of a higher daily dose of tamsulosin (0.8mg) on stent-related symptoms. The objective of this study is to assess two different dosing regimens (0.4 mg QD vs. 0.4 mg BID) of tamsulosin for ureteral stent-related discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 70 years old.
* Planning to undergo ureteroscopy with ureteral stent placement at our site.
* Able to read and understand an English language survey (USSQ).

Exclusion Criteria:

1. Patients who are unable to provide informed consent.
2. Patients who are already taking an alpha-blocker.
3. Patients with hypersensitivity or known adverse side effects of tamsulosin or its ingredients and those who are not candidates for tamsulosin per attending Urologist discretion.
4. Patients with a preexisting bladder condition including UTI within 30 days of the procedure.
5. Patients with hepatitis C on boceprevir.
6. Patients who have medical conditions known to be associated with chronic pain, those taking medications for chronic pain such as gabapentin or a chronic opioid per the judgement of the PI, or those with a pain contract on file.
7. Women who are pregnant or planning to become pregnant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-02-18 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Ureteric Stent Symptoms Questionnaire | 1 week post-stent placement
  Scales for each question are 1 to 5, with 5 indicated more severe symptoms. Subscale scores are the sum of all questions included in the subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Ferroni, MD, Principal Investigator — Gundersen Health System
Locations (1):
- Gundersen Health System, La Crosse, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koprowski C, Kim C, Modi PK, Elsamra SE. Ureteral Stent-Associated Pain: A Review. J Endourol. 2016 Jul;30(7):744-53. doi: 10.1089/end.2016.0129. Epub 2016 May 23. PMID 27125392
- [Background] Bosio A, Alessandria E, Dalmasso E, Peretti D, Agosti S, Bisconti A, Destefanis P, Passera R, Gontero P. How bothersome double-J ureteral stents are after semirigid and flexible ureteroscopy: a prospective single-institution observational study. World J Urol. 2019 Jan;37(1):201-207. doi: 10.1007/s00345-018-2376-6. Epub 2018 Jun 19. PMID 29923014
- [Background] Joshi HB, Newns N, Stainthorpe A, MacDonagh RP, Keeley FX Jr, Timoney AG. Ureteral stent symptom questionnaire: development and validation of a multidimensional quality of life measure. J Urol. 2003 Mar;169(3):1060-4. doi: 10.1097/01.ju.0000049198.53424.1d. PMID 12576846
- [Background] Lamb AD, Vowler SL, Johnston R, Dunn N, Wiseman OJ. Meta-analysis showing the beneficial effect of alpha-blockers on ureteric stent discomfort. BJU Int. 2011 Dec;108(11):1894-902. doi: 10.1111/j.1464-410X.2011.10170.x. Epub 2011 Mar 31. PMID 21453351
- [Background] Dellis AE, Papatsoris AG, Keeley FX Jr, Bamias A, Deliveliotis C, Skolarikos AA. Tamsulosin, Solifenacin, and Their Combination for the Treatment of Stent-Related Symptoms: A Randomized Controlled Study. J Endourol. 2017 Jan;31(1):100-109. doi: 10.1089/end.2016.0663. Epub 2016 Nov 29. PMID 27809592